CLINICAL TRIAL: NCT02067988
Title: Adjuvant Hepatic Holmium-166-radioembolization in Patients With Unresectable Liver Metastases of Neuroendocrine Origin, Who Have Been Treated With Lutetium-177-dotatate
Brief Title: Holmium-166-radioembolization in NET After Lutetium-177-dotatate; an Efficacy Study
Acronym: HEPAR_Plus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Marnix Lam, MD, PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL45329.041.13
Record Dates: First submitted 2014-02-13; First posted 2014-02-20 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Neuroendocrine Tumors
Keywords: Radioembolization; Somatostatin receptor treatment; Neuroendocrine tumors; Liver metastases
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Holmium-166 microspheres hepatic radioembolization, adjuvant to systemic 177Lu-dotatate.
  Interventions: Device: Holmium-166 microspheres hepatic radioembolization.

INTERVENTIONS:
Device: Holmium-166 microspheres hepatic radioembolization. — Holmium-166 microspheres hepatic radioembolization.

SUMMARY:
Patients with gastroenteropancreatic neuroendocrine tumours (NET) often die from intrahepatic disease or are excluded from liver-directed treatment because of extrahepatic disease. Adjuvant liver-directed treatment is warranted to control both intra- and extrahepatic disease. Patients with liver metastases of NET will be included in this study (n = 30-48).The efficacy and toxicity of adjuvant 166Ho-radioembolization (166Ho-RE) after systemic 177Lu-dotatate will be studied in a non-comparative phase II study. The study is an interventional, treatment, non-randomized, open label, non-comparative, phase II study. 166Ho-RE will be performed via a catheter during angiography.

DETAILED DESCRIPTION:
Acronym :

Holmium Embolization Particles for Arterial Radiotherapy Plus 177Lu-dotatate in Salvage NET patients- HEPAR PLUS-trial.

Rationale:

Patients with gastroenteropancreatic neuroendocrine tumours (NET) often die from intrahepatic disease or are excluded from liver-directed treatment because of extrahepatic disease. Adjuvant liver-directed treatment is warranted to control both intra- and extrahepatic disease.

Objective:

Primary objectives:

* To evaluate efficacy of adjuvant 166Ho-radioembolization (166Ho-RE) after systemic 177Lu-dotatate in a non-comparative phase II study.
* To establish the safety and toxicity profile of adjuvant 166Ho-RE after systemic treatment with 177Lu-dotatate.

Secondary objectives:

* To evaluate Quality of Life (QoL).
* To evaluate biodistribution / dosimetry.

Study design:

Interventional, treatment, non-randomized, open label, non-comparative, phase II study.

Study population:

Patients with liver metastases of NET will be included in this study (n = 30-48). These male and female patients must be aged ≥18 years. All NET histologies are acceptable, provided no standard therapeutic options are available, such as chemotherapy and surgery.

Intervention:

166Ho-RE will be performed via a catheter during angiography.

Study endpoints:

Primary endpoints:

* Tumour response at 3 months.
* Safety and toxicity profile of 166Ho-RE as adjuvant treatment after 177Lu-dotatate.

Secondary endpoints:

* Changes in tumour markers.
* Quality of Life (QoL).
* Biodistribution / Dosimetry.

Duration of treatment:

The study consists of a screening phase of approximately 2 weeks followed by a treatment phase of approximately 2-3 weeks. Patients will be followed until liver specific tumour progression or death has occurred, to a maximum of 12 months.

Methodology:

A first cohort of 30 patients will be treated with 166Ho-RE. After the first cohort, up to 3 additional cohorts of 6 patients will be treated with 166Ho-RE. The total number of patients treated in the HEPAR PLUS trial will therefore be at least 30 and at most 48 patients, depending on the observed number of responses. Early termination at a response interim analysis (after 30, 36 or 42 patients) is determined by pre-defined boundaries on the number of observed responses. The boundary in favour of treatment effect may be crossed before 30 patients are reached, but then the study will continue to at least 30 patients to allow estimation of the key secondary endpoints.

Number of study centers:

Single center (UMC Utrecht).

Adverse events:

All adverse events will be recorded throughout the study.

Inclusion period:

January 2014 - January 2017

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have given written informed consent.
2. Female or male aged 18 years and over.
3. Confirmed histological diagnosis NET, including bronchial carcinoids, and metastatic malignancy with liver metastases without standard therapeutic options for treatment including chemotherapy or surgery.
4. Patients must have been treated with 4 cycles of 200 mCi 177Lu-dotatate, the last cycle within 8-12 weeks of 166Ho-RE.
5. Life expectancy of 12 weeks or longer.
6. World Health Organisation (WHO) Performance status 0-2.
7. Liver disease with three or more measurable liver lesions according to the RECIST 1.1 criteria.
8. Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

1. Brain metastases or spinal cord compression, unless irradiated at least 4 weeks prior to the date of the experimental treatment and stable without steroid treatment for at least 1 week.
2. Radiation therapy within the last 4 weeks before the start of study therapy.
3. The last dose of prior chemotherapy has been received less than 4 weeks prior the start of study therapy.
4. Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy.
5. Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events grade 2 from previous anti-cancer therapy.
6. Serum bilirubin > 1.5 x Upper Limit of Normal (ULN).
7. Glomerular filtration rate <35 ml/min, determined according to the Modification of Diet in Renal Disease formula.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) > 5 x ULN.
9. Leukocytes < 3.0 x 109/l and/or platelet count < 100 x 109/l.
10. Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
11. Pregnancy or nursing (women of child-bearing potential).
12. Patients suffering from diseases with an increased chance of liver toxicity.
13. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
14. Patients who are declared incompetent.
15. Previous enrolment in the present study or previous treatment with RE.
16. Female patients who are not using an acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) OR are less than 1 year postmenopausal or surgically sterile during their participation in this study (from the time they sign the consent form) to prevent pregnancy.
17. Male patients who are not surgically sterile or do not use an acceptable method of contraception during their participation in this study (from the time they sign the consent form) to prevent pregnancy in a partner.
18. Patients with abnormalities of the bile ducts (such as stents) with an increased chance of infections of the bile ducts (papillotomy and cholecystectomy are allowed). Or evidence of extensive portal hypertension, splenomegaly, ascites or active hepatitis (B and/or C).
19. Body weight over 150 kg.
20. Severe allergy for i.v. contrast (Visipaque®), used for CT evaluation, pre-treatment angiography and treatment angiography.
21. Liver tumour involvement ≥70% as quantified on CT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-02; Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Response (RECIST 1.1 Partial plus complete) | 3 months
  To evaluate efficacy of adjuvant 166Ho-radioembolization (166Ho-RE) after systemic 177Lu-dotatate in a non-comparative phase II study

SECONDARY OUTCOMES:
Quality of Life (QoL) | 3 months
  To evaluate QoL using EORTC questionnaire. The impact of treatment on QoL will be compared to tumour response, and other parameters. A questionnaire in the patient's native language will be provided.
Biodistribution | 3 months
  To evaluate biodistribution using CT and quantitative SPECT.
Dosimetry | 3 months
  To evaluate dosimetry using CT and quantitative SPECT. The imaging protocol after injection of 166Ho-PLLA-MS will consist of a dual isotope fusion SPECT/CT protocol.
AD Adverse events | 1 year
  To establish the safety and toxicity profile of treatment with 166Ho-microspheres as an adjuvant treatment after 177Lu-dotatate. This profile will be established using CTCAE (incl. SAE) methodology (CTCAE version 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Marnix G Lam, MD, PhD, Principal Investigator — UMC Utrecht, The Netherlands
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Stella M, van Rooij R, Lam MGEH, de Jong HWAM, Braat AJAT. Automatic healthy liver segmentation for holmium-166 radioembolization dosimetry. EJNMMI Res. 2023 Jul 15;13(1):68. doi: 10.1186/s13550-023-00996-1. PMID 37453996
- [Derived] Stella M, Braat AJAT, Lam MGEH, de Jong HWAM, van Rooij R. 166Holmium-99mTechnetium dual-isotope imaging: scatter compensation and automatic healthy-liver segmentation for 166Holmium radioembolization dosimetry. EJNMMI Phys. 2022 Apr 21;9(1):30. doi: 10.1186/s40658-022-00459-x. PMID 35445948
- [Derived] Ebbers SC, Brabander T, Tesselaar MET, Hofland J, Braat MNGJA, Wessels FJ, Barentsz MW, Lam MGEH, Braat AJAT. Inflammatory markers and long term hematotoxicity of holmium-166-radioembolization in liver-dominant metastatic neuroendocrine tumors after initial peptide receptor radionuclide therapy. EJNMMI Res. 2022 Feb 2;12(1):7. doi: 10.1186/s13550-022-00880-4. PMID 35107642
- [Derived] Stella M, Braat A, Lam M, de Jong H, van Rooij R. Quantitative 166Ho-microspheres SPECT derived from a dual-isotope acquisition with 99mTc-colloid is clinically feasible. EJNMMI Phys. 2020 Jul 14;7(1):48. doi: 10.1186/s40658-020-00317-8. PMID 32666401
- [Derived] Braat AJAT, Bruijnen RCG, van Rooij R, Braat MNGJA, Wessels FJ, van Leeuwaarde RS, van Treijen MJC, de Herder WW, Hofland J, Tesselaar MET, de Jong HWAM, Lam MGEH. Additional holmium-166 radioembolisation after lutetium-177-dotatate in patients with neuroendocrine tumour liver metastases (HEPAR PLuS): a single-centre, single-arm, open-label, phase 2 study. Lancet Oncol. 2020 Apr;21(4):561-570. doi: 10.1016/S1470-2045(20)30027-9. Epub 2020 Feb 26. PMID 32112737
- [Derived] Braat AJAT, Kwekkeboom DJ, Kam BLR, Teunissen JJM, de Herder WW, Dreijerink KMA, van Rooij R, Krijger GC, de Jong HWAM, van den Bosch MAAJ, Lam MGEH. Additional hepatic 166Ho-radioembolization in patients with neuroendocrine tumours treated with 177Lu-DOTATATE; a single center, interventional, non-randomized, non-comparative, open label, phase II study (HEPAR PLUS trial). BMC Gastroenterol. 2018 Jun 15;18(1):84. doi: 10.1186/s12876-018-0817-8. PMID 29902988